CLINICAL TRIAL: NCT02937818
Title: A Phase II, Open-Label, Multi-Arm Study to Determine the Preliminary Efficacy of Novel Combinations of Treatment in Patients With Platinum Refractory Extensive-Stage Small-Cell Lung Cancer
Brief Title: A Phase II, Study to Determine the Preliminary Efficacy of Novel Combinations of Treatment in Patients With Platinum Refractory Extensive-Stage Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419QC00002; 2016-001202-42 (EudraCT Number)
Record Dates: First submitted 2016-10-05; First posted 2016-10-19 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Platinum Refractory Extensive-Stage Small Cell Lung Carcinoma
Keywords: Platinum Refractory Extensive-Stage Carcinoma, Small Cell Lung; Platinum Refractory Extensive-Stage Oat Cell Carcinoma of Lung; Platinum Refractory Extensive-Stage Oat Cell Lung Cancer; Platinum Refractory Extensive-Stage Small Cell Cancer Of The Lung; Platinum Refractory Extensive-Stage Small Cell Lung Cancer
MeSH Terms: interventions — durvalumab; tremelimumab; adavosertib; Carboplatin; ceralasertib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARM A (Experimental)
  Interventions: Drug: Durvalumab and Tremelimumab
- ARM B (Experimental)
  Interventions: Drug: AZD1775 and carboplatin (CBPT)
- ARM C (Experimental)
  Interventions: Drug: AZD6738 and olaparib

INTERVENTIONS:
Drug: Durvalumab and Tremelimumab — Durvalumab + tremelimumab via intravenous (IV) infusion every 4 weeks (q4w), starting on Week 0, for up to a total of 4 months (4 cycles) followed by durvalumab monotherapy via IV infusion q4w, starting on Week 16 until PD, or for other discontinuation criteria.
  Arms: ARM A
Drug: AZD1775 and carboplatin (CBPT) — AZD1775 twice daily (oral) for 2.5 days from Day 1 + CBDP area under the curve 5 (Day1) (IV); every 3 weeks.
  Arms: ARM B
Drug: AZD6738 and olaparib — AZD6738 once a day (oral) for 7 days from Day 1 + olaparib twice a day(oral) for 28 days from Day 1, every 4 weeks
  Arms: ARM C

SUMMARY:
Study design This is a Phase II, open-label, multi-drug, multi-center, multi-arm, signal-searching study in patients with extensive-stage small-cell lung cancer (SCLC) who have refractory or resistant disease from prior platinum-based chemotherapy.

DETAILED DESCRIPTION:
This study is modular in design, allowing evaluation of the preliminary efficacy, safety, tolerability, and immunogenicity of novel combinations of immunotherapies and/or deoxyribonucleic acid (DNA) damage repair inhibitors in patients with platinum refractory or resistant extensive-stage-disease SCLC. Patients who have progressive disease (PD) during first-line platinum-based chemotherapy (platinum refractory) or PD within 90 days after completing first-line platinum-based chemotherapy (platinum resistant) will be enrolled to the study. The primary objective of the study is to assess the preliminary efficacy of each treatment arm based on objective response rate (ORR).

This study consists of a number of arms (sub-studies), each evaluating the efficacy, safety, and tolerability of a specific agent or combination. This study was initially open with 2 arms (Arms A and B), and additional arms may open, provided there is compelling rationale for the combination and safe and tolerable doses and schedules have been determined from ongoing Phase I studies. There are 2 pre-defined arms:

A. Durvalumab + tremelimumab followed by durvalumab monotherapy B. AZD1775 + carboplatin (CBDP)

Further arm was added in amendment 3:

C. AZD6738 + olaparib Amendment #4 was updated with possibility to allow expansion of any arm, to a total of 40 eligible subjects, based on Review Committee assessment of data from the first 20 subjects (from Stage 1 and Stage 2). Currently Arm A will enroll 20 additional patients into expansion.

ELIGIBILITY:
Inclusion criteria (applicable to all arms)

* Adults with histologically or cytologically documented ED SCLC who have demonstrated progressive disease either during first-line platinum-based chemotherapy (platinum refractory) or within 90 days of completing platinum based-chemotherapy (platinum resistant) and have not received further treatment.
* Brain metastases must be asymptomatic or treated and stable off steroids and anti-convulsants for at least 1 month prior to study treatment.
* At least 1 lesion, not previously irradiated, that can be accurately measured at baseline (per RECIST v 1.1 guidelines)
* Life expectancy of at least 8 weeks.
* WHO/ ECOG PS of 0-1 at enrollment.

Inclusion criteria (Arm A specific)

* Body weight >30 kg.
* No prior exposure to immune mediated therapy, excluding therapeutic anticancer vaccines.

Inclusion criteria (Arm B specific) • Able and willing to swallow oral medication.

Inclusion criteria (Arm C specific)

• Able and willing to swallow oral medication.

Exclusion criteria (applicable to all arms):

* Participation in another clinical study, major surgery, radiation therapy within 28 days.
* Any condition that, in the opinion of the Investigator, would interfere with the evaluation of the IP or interpretation of patient safety or study results.
* Uncontrolled intercurrent illness, including but not limited to interstitial lung disease.
* History of another primary malignancy, leptomeningeal carcinomatosis or spinal cord compression.

Exclusion criteria (Arm A specific)

* Active autoimmune disease, including a paraneoplastic syndrome.
* Active or prior documented autoimmune or inflammatory disorders.
* Any unresolved toxicity (CTCAE Grade >2) from previous anticancer therapy.
* Active infection including tuberculosis, HIV, Hepatitis B or C.

Exclusion criteria (Arm B specific)

* Prior exposure to any WEE1 inhibitors.
* Products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4. Co-administration of rosuvastatin, atorvastatin, simvastatin and lovastatin, aprepitant or fosaprepitant or any herbal preparations. Grapefruit and Seville oranges should be avoided while taking AZD1775.
* Any known hypersensitivity or contraindication to IP or CBDP.
* QTcF > 470 msec or congenital long QT syndrome.
* Any current or within 6 months cardiac diseases NYHA ≥ Class 2: unstable angina pectoris, congestive heart failure, acute MI, conduction abnormality not controlled with pacemaker or medication, significant ventricular or supraventricular arrhythmias.
* A recent history of Torsades de pointes.

Exclusion criteria (Arm C specific)

* Cytotoxic chemotherapy within 21 days of Cycle 1 Day 1 is not permitted
* Previous treatment with a PARP inhibitor (including olaparib) or ATR inhibitor
* Concomitant use of known strong CYP3A inhibitors and moderate CYP3A inhibitors
* Concomitant use of known strong and moderate CYP3A inducers
* Persisting (> 4 weeks) severe pancytopenia due to previous therapy
* Cardiac dysfunction
* Refractory nausea and vomitting, chronic gastrointenstinal diseases or previous significant bowel resection
* Patients with uncontrolled seizures
* Intenstinal obstruction or CTCAE grade 3 or grade 4 GI bleeding within 4 weeks before dosing

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haiyi Jiang, M.D., Study Director — AstraZeneca
Locations (12):
- Research Site, Gauting, Germany
- Hungary (4):
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
- Poland (2):
  - Research Site, Poznan
  - Research Site, Warsaw
- Spain (2):
  - Research Site, Seville
  - Research Site, Valencia
- Ukraine (3):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Sumy

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00002&attachmentIdentifier=e9bf5453-5908-48cd-8e57-c658c9e5ff5b&fileName=D419QC00002_CSP_redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00002&attachmentIdentifier=4efd214e-ac11-406a-a7ef-db809ed51fda&fileName=D419QC00002_SAP_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419QC00002&attachmentIdentifier=41707687-adcb-45ce-a908-85b066378e8d&fileName=D419QC00002_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 28-Nov-2016 and 22-Jun-2020, at 11 study centers in 5 countries (Germany, Hungary, Poland, Spain, and Ukraine).
Pre-assignment Details: Participants who met the inclusion exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
Groups:
- Arm A: Durvalumab + Tremelimumab (Original Cohort): Participants received durvalumab 1500 mg + tremelimumab 75 mg via intravenous (IV) infusion every 4 weeks (q4w), starting on Week 0, for up to a total of 4 months (4 cycles) followed by durvalumab monotherapy 1500 mg via IV infusion q4w, starting on Week 16 until confirmed progressive disease (PD), or other discontinuation criteria.
- Arm A: Durvalumab + Tremelimumab (Expansion Cohort): Participants received durvalumab 1500 mg + tremelimumab 75 mg via intravenous (IV) infusion every 4 weeks (q4w), starting on Week 0, for up to a total of 4 months (4 cycles) followed by durvalumab monotherapy 1500 mg via IV infusion q4w, starting on Week 16 until confirmed PD, or other discontinuation criteria.
- Arm B: Adavosertib + Carboplatin: Participants orally received adavosertib 225 mg twice daily (BID) for 2.5 days from Day 1 + carboplatin area under the curve (AUC) 5 Day 1 IV, every 3 weeks (q3w).
- Arm C: Ceralasertib (AZD6738) + Olaparib: Participants orally received ceralasertib 160 mg once daily (QD) Days 1 to 7 + olaparib 300 mg BID Days 1 to 28, q4w.
Period: Overall Study
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) | Arm B: Adavosertib + Carboplatin | Arm C: Ceralasertib (AZD6738) + Olaparib
Started | 21 | 20 | 10 | 21
Completed | 0 | 0 | 0 | 0
Not Completed | 21 | 20 | 10 | 21
Not completed — Participants decision | 2 | 1 | 1 | 1
Not completed — Adverse Event | 2 | 4 | 1 | 1
Not completed — Disease progression | 17 | 15 | 7 | 19
Not completed — Condition under investigation worsened | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) | Arm B: Adavosertib + Carboplatin | Arm C: Ceralasertib (AZD6738) + Olaparib | Total
Number analyzed (Participants) | 21 | 20 | 10 | 21 | 72
Age, Customized [Count of Participants; unit: Participants]
  < 50 | 2 | 0 | 1 | 2 | 5
  ≥ 50 to < 65 | 13 | 12 | 5 | 12 | 42
  ≥ 65 to < 75 | 6 | 6 | 3 | 5 | 20
  ≥ 75 to < 80 | 0 | 2 | 1 | 2 | 5
  ≥ 80 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 2 | 7 | 19
  Male | 15 | 16 | 8 | 14 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 21 | 19 | 10 | 21 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 21 | 20 | 10 | 21 | 72
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Overall Response Rate (ORR) using Investigator assessments according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. ORR was defined as the number (percentage) of participants with a confirmed Complete Response (CR) or confirmed Partial Response (PR) and was estimated for each treatment arm with corresponding 2-sided 95% exact confidence intervals (CIs). A confirmed response of CR/PR meant that a response of CR/PR was recorded at one visit and confirmed by repeat imaging, preferably at the next regularly scheduled imaging visit, and not less than 4 weeks after the visit when the response was first observed, with no evidence of progression between the initial and CR/PR confirmation visit.
Time Frame: Until disease progression [PD] (Up to 3.5 Years)
Population: The FAS included all treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) | Arm B: Adavosertib + Carboplatin | Arm C: Ceralasertib (AZD6738) + Olaparib
Number analyzed (Participants) | 21 | 20 | 10 | 21
Participants | 2 | 1 | 0 | 1

2. Secondary Outcome: Duration of Response (DoR)
Description: The DoR was defined as the time from the date of first documented response (which was subsequently confirmed) CR/PR until the date of documented progression, or death in the absence of disease progression. The DoR in participants with confirmed objective response are reported.
Time Frame: Until disease progression or data cut-off or Death (Up to 3.5 Years)
Population: The FAS included all treated participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) | Arm B: Adavosertib + Carboplatin | Arm C: Ceralasertib (AZD6738) + Olaparib
Number analyzed (Participants) | 2 | 1 | 0 | 1
Months | NA [1.5 to NA] — Objective response not reached | 3 [3 to 3] |  | 8.5 [8.5 to 8.5]

3. Secondary Outcome: Percentage of Participants With Disease Control at 12 Weeks
Description: The disease control rate (DCR) at 12 weeks was defined as the percentage of participants who had a best objective response of CR or PR in the first 13 weeks or who had demonstrated stable disease (SD) for a minimum interval of 11 weeks following the start of study treatment. The DCR was determined programmatically based on RECIST 1.1 using site Investigator data and all data up until the first progression event.
Time Frame: At 12 Weeks
Population: The FAS included all treated participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) | Arm B: Adavosertib + Carboplatin | Arm C: Ceralasertib (AZD6738) + Olaparib
Number analyzed (Participants) | 21 | 20 | 10 | 21
Percentage of Participants | 38.1 | 15.0 | 30.0 | 38.1

4. Secondary Outcome: Time to Response (TTR)
Description: The TTR (per RECIST 1.1 as assessed by the Investigator) was defined as the time from the date of first dose until the first date of documented response.
Time Frame: Until disease progression or data cut-off or Death (Up to 3.5 Years)
Population: The FAS included all treated participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) | Arm B: Adavosertib + Carboplatin | Arm C: Ceralasertib (AZD6738) + Olaparib
Number analyzed (Participants) | 2 | 1 | 0 | 1
Months | 1.8 [1.7 to 1.8] | 1.8 [1.8 to 1.8] |  | 1.7 [1.7 to 1.7]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: The PFS (per RECIST 1.1 according to the Investigator's assessment) was defined as the time from the date of the first dose of study treatment until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdrew from allocated therapy or received another anti-cancer therapy prior to progression.
Time Frame: Until disease progression or data cut-off or Death (Up to 3.5 Years)
Population: The FAS included all treated participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) | Arm B: Adavosertib + Carboplatin | Arm C: Ceralasertib (AZD6738) + Olaparib
Number analyzed (Participants) | 21 | 20 | 10 | 21
Months | 1.91 [1.77 to 4.34] | 1.77 [1.02 to 2.20] | 2.60 [0.56 to 4.83] | 2.92 [1.81 to 4.53]

6. Secondary Outcome: Overall Survival (OS)
Description: The OS was defined as the time from the date of the first dose of study treatment until death due to any cause.
Time Frame: Until disease progression or data cut-off or Death (Up to 3.5 Years)
Population: The FAS included all treated participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) | Arm B: Adavosertib + Carboplatin | Arm C: Ceralasertib (AZD6738) + Olaparib
Number analyzed (Participants) | 21 | 20 | 10 | 21
Months | 5.95 [1.91 to 10.61] | 3.37 [1.91 to 7.66] | 4.67 [0.56 to 5.98] | 7.56 [4.21 to 12.58]

7. Secondary Outcome: Time to Maximum Concentration (Tmax)
Description: Time to maximum concentration for ceralasertib and olaparib are reported.
Time Frame: Cycle 1 (each cycle was 28 days in length) Day 1 (post-dose)
Population: Pharmacokinetic Analysis Set: all participants who received at least 1 dose of study treatment and had post-dose data available, excluding those who had a deviation considered by the sponsor to have a potential impact on the interpretation of the pharmacokinetic analyses.
Measure: Median (Full Range); unit: Hour
Groups:
- Ceralasertib (AZD6738); Olaparib: Participants orally received ceralasertib 160 mg once daily (QD) Days 1 to 7 + olaparib 300 mg BID Days 1 to 28, q4w.
Arm/Group | Ceralasertib (AZD6738) | Olaparib
Number analyzed (Participants) | 21 | 21
Hour | 1.250 [1.00 to 6.08] | 1.800 [1.00 to 6.08]

8. Secondary Outcome: Maximum Concentration (Cmax)
Description: Maximum concentration for ceralasertib and olaparib are reported.
Time Frame: Cycle 1 (each cycle was 28 days in length) Day 1 (post-dose)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ceralasertib (AZD6738) | Olaparib
Number analyzed (Participants) | 21 | 21
µg/mL | 4.215 (27.7129) | 6.558 (39.9411)

9. Secondary Outcome: Partial Area Under the Concentration-time Curve (AUC0-6)
Description: Partial area under the concentration-time curve for ceralasertib and olaparib are reported.
Time Frame: Cycle 1 (each cycle was 28 days in length) Day 1 (post-dose) and Cycle 1 Day 7 (pre-dose and post-dose)
Population: Pharmacokinetic Analysis Set: all participants who received at least 1 dose of study treatment and had post-dose data available, excluding those who had a deviation considered by the sponsor to have a potential impact on the interpretation of the pharmacokinetic analyses. Here, number analyzed in each row signifies only participants with available data that were analyzed for that specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Ceralasertib (AZD6738) | Olaparib
Number analyzed (Participants) | 20 | 21
h*µg/mL
  Cycle 1, Day 1 | 18.346 (34.6952) | 26.356 (42.2963)
  Cycle 1, Day 7: number analyzed (Participants) | 10 | 10
  Cycle 1, Day 7 | 23.666 (23.9202) | 42.016 (33.7599)

10. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC0-t)
Description: Area under the concentration-time curve from time zero to the last measurable concentration for Ceralasertib and Olaparib are reported.
Time Frame: Cycle 1 (each cycle was 28 days in length) Day 1 (post-dose) and Cycle 1 Day 7 (pre-dose and post-dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Ceralasertib (AZD6738) | Olaparib
Number analyzed (Participants) | 21 | 21
h*µg/mL
  Cycle 1, Day 1 | 18.575 (34.5074) | 26.973 (41.4461)
  Cycle 1, Day 7: number analyzed (Participants) | 10 | 10
  Cycle 1, Day 7 | 24.061 (23.0923) | 62.535 (42.4552)

11. Secondary Outcome: Time to Maximum Concentration at Steady State (Tmax,ss)
Description: Time to maximum concentration at steady state for Ceralasertib and Olaparib are reported.
Time Frame: Cycle 1 (each cycle was 28 days in length) Day 7 (pre-dose and post-dose)
Population: as for outcome 7
Measure: Median (Full Range); unit: Hour
Arm/Group | Ceralasertib (AZD6738) | Olaparib
Number analyzed (Participants) | 10 | 10
Hour | 1.875 [0.63 to 6.08] | 2.708 [0.63 to 4.50]

12. Secondary Outcome: Maximum Concentration at Steady State (Cmax,ss)
Description: Maximum concentration at steady state for Ceralasertib and Olaparib are reported.
Time Frame: Cycle 1 (each cycle was 28 days in length) Day 7 (pre-dose and post-dose)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ceralasertib (AZD6738) | Olaparib
Number analyzed (Participants) | 10 | 10
µg/mL | 5.176 (23.4058) | 9.189 (30.4888)

13. Secondary Outcome: Minimum Concentration at Steady State (Cmin,ss)
Description: Minimum concentration at steady state for Ceralasertib and Olaparib are reported.
Time Frame: Cycle 1 (each cycle was 28 days in length) Day 7 (pre-dose and post-dose)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Ceralasertib (AZD6738) | Olaparib
Number analyzed (Participants) | 10 | 10
µg/mL | 1.119 (55.9070) | 2.376 (61.8191)

14. Secondary Outcome: Area Under the Concentration-time Curve at Steady State (AUCss)
Description: Area under the concentration-time curve at steady state at steady state for Ceralasertib and Olaparib are reported.
Time Frame: Cycle 1 (each cycle was 28 days in length) Day 7 (pre-dose and post-dose)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Ceralasertib (AZD6738) | Olaparib
Number analyzed (Participants) | 10 | 9
h*µg/mL | NA (NA) — There were not enough pharmacokinetic data points collected to calculate AUCss | 67.929 (37.4297)

15. Secondary Outcome: Apparent Clearance of Drug at Steady State at Steady State (CLss/F)
Description: Area under the concentration-time curve at steady state at steady state for Ceralasertib and Olaparib are reported.
Time Frame: Cycle 1 (each cycle was 28 days in length) Day 7 (pre-dose and post-dose)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre/hour
Arm/Group | Ceralasertib (AZD6738) | Olaparib
Number analyzed (Participants) | 10 | 9
Litre/hour | NA (NA) — There were not enough pharmacokinetic data points collected to calculate CLss/F | 4.416 (42.3171)

16. Secondary Outcome: Serum Concentrations of Durvalumab and Tremelimumab
Description: Serum concentrations of Durvalumab and Tremelimumab are reported.
Time Frame: Durvalumab: Cycle 1 (each cycle was 4 weeks) Day 1(post-dose); Cycle 2 Day 1(pre-dose); Cycle 5 Day 1 (pre-dose); Tremelimumab: Cycle 1 (each cycle was 4 weeks) Day 1 (post-dose); Cycle 2 Day 1 (pre-dose); Cycle 5 Day 1 (No dose); Cycle 7 Day 1 (No dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort)
Number analyzed (Participants) | 21
μg/mL
  Durvalumab: Cycle 1 Day 1 (Post-dose) | 391.192 (23.5990)
  Durvalumab: Cycle 2 Day 1 (Pre-dose): number analyzed (Participants) | 17
  Durvalumab: Cycle 2 Day 1 (Pre-dose) | 55.590 (53.0745)
  Durvalumab: Cycle 5 Day 1 (Pre-dose): number analyzed (Participants) | 7
  Durvalumab: Cycle 5 Day 1 (Pre-dose) | 116.846 (51.0036)
  Tremelimumab: Cycle 1 Day 1 (Post-dose) | 18.299 (20.8181)
  Tremelimumab: Cycle 2 Day 1 (Pre-dose): number analyzed (Participants) | 16
  Tremelimumab: Cycle 2 Day 1 (Pre-dose) | 2.650 (53.1007)
  Tremelimumab: Cycle 5 Day 1 (No dose): number analyzed (Participants) | 6
  Tremelimumab: Cycle 5 Day 1 (No dose) | 5.005 (38.3784)
  Tremelimumab: Cycle 7 Day 1 (No dose): number analyzed (Participants) | 3
  Tremelimumab: Cycle 7 Day 1 (No dose) | 0.784 (66.3469)

17. Secondary Outcome: Plasma Concentrations of Adavosertib and Carboplatin
Description: Plasma concentrations of Adavosertib and Carboplatin are reported.
Time Frame: Adavosertib: Cycle 1 (each cycle was 21 days) Day 3 (pre-dose and post-dose); Cycle 3 Day 3 (pre-dose and post-dose); Carboplatin: Cycle 1 (each cycle was 21 days) Day 1 (post-dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Arm B: Adavosertib + Carboplatin
Number analyzed (Participants) | 10
nM
  Adavosertib: Cycle 1 Day 3 (Pre-dose): number analyzed (Participants) | 9
  Adavosertib: Cycle 1 Day 3 (Pre-dose) | 551.489 (41.5823)
  Adavosertib: Cycle 1 Day 3 (Post-dose): number analyzed (Participants) | 9
  Adavosertib: Cycle 1 Day 3 (Post-dose) | 728.342 (62.3968)
  Adavosertib: Cycle 3 Day 3 (Pre-dose): number analyzed (Participants) | 4
  Adavosertib: Cycle 3 Day 3 (Pre-dose) | 606.571 (46.7716)
  Adavosertib: Cycle 3 Day 3 (Post-dose): number analyzed (Participants) | 3
  Adavosertib: Cycle 3 Day 3 (Post-dose) | 805.270 (68.0275)
  Carboplatin: Cycle 1 Day 1 (Post-dose) | 12834.615 (27.5493)

18. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. SAE is an AE that results in any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, or is a significant medical event.
Time Frame: Day 1 until disease progression, and follow-up visit (Up to 3.5 Years)
Population: The FAS included all treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) | Arm B: Adavosertib + Carboplatin | Arm C: Ceralasertib (AZD6738) + Olaparib
Number analyzed (Participants) | 21 | 20 | 10 | 21
Participants
  Any AE | 16 | 17 | 8 | 18
  Any AE causally related to any study treatment | 10 | 9 | 8 | 16
  Any AE with outcome = death | 1 | 0 | 1 | 1
  Any SAE | 6 | 8 | 4 | 7
  Any AE leading to discontinuation of any study treatment | 2 | 4 | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 1 until disease progression, and follow-up visit (Up to 3.5 Years)
Arm/Group | Arm A: Durvalumab + Tremelimumab (Original Cohort) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) | Arm B: Adavosertib + Carboplatin | Arm C: Ceralasertib (AZD6738) + Olaparib
All-Cause Mortality (participants affected / at risk) | 19/21 | 16/20 | 10/10 | 15/21
Serious Adverse Events (participants affected / at risk) | 6/21 | 8/20 | 4/10 | 7/21
Other Adverse Events (participants affected / at risk) | 14/21 | 16/20 | 8/10 | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Durvalumab + Tremelimumab (Original Cohort) (N=21) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) (N=20) | Arm B: Adavosertib + Carboplatin (N=10) | Arm C: Ceralasertib (AZD6738) + Olaparib (N=21)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (3) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematotoxicity (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Durvalumab + Tremelimumab (Original Cohort) (N=21) | Arm A: Durvalumab + Tremelimumab (Expansion Cohort) (N=20) | Arm B: Adavosertib + Carboplatin (N=10) | Arm C: Ceralasertib (AZD6738) + Olaparib (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 3 (5) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 7 (14) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 5 (6) | 1 (1) | 3 (6) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (3) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2) | 3 (6) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 6 (13) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 7 (13) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 3 (13) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 3 (6) | 3 (4)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0) | 1 (3) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Influenza (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results are Sponsor's intellectual property and PIs cannot present or publish results without prior Sponsor approval.

DOCUMENTS (2):
  • Study Protocol (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT02937818/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT02937818/SAP_001.pdf